CLINICAL TRIAL: NCT00655564
Title: Long-Term One Year Use of Alefacept (Amevive®) in Moderate to Severe Chronic Plaque Type Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00004816; 32547 Contract number
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alefacept (Experimental): Alefacept's FDA indication is for the treatment of adult subjects with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy. The approved dosing regimen is 15mg once weekly as an intramuscular injection or 7.5mg given once weekly as an intravenous bolus. The recommended regimen is a course of 12 weeks.
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — Alefacept's FDA indication is for the treatment of adult subjects with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy. The approved dosing regimen is 15mg once weekly as an intramuscular injection or 7.5mg given once weekly as an intravenous bolus. The recommended regimen is a course of 12 weeks.
  Alefacept is supplied as a lyophilized powder. Alefacept contains LFA3-IgG1 Fusion Protein and excipient materials (citrate, glycine and sucrose).
  Other Names: Amevive®

SUMMARY:
The purpose of this research study is to see how well the medication Alefacept (Amevive®) works for continuous treatment of chronic plaque psoriasis. The US Food and Drug Administration (FDA) has approved Alefacept in an intermittent dosage schedule of 15 mg weekly injection for 12 weeks followed by 12 weeks off treatment.

DETAILED DESCRIPTION:
To estimate the efficacy of continuous use of alefacept (15mg IM/week) in the treatment of moderate to severe chronic plaque type psoriasis as defined as Investigator Global Assessment (IGA) of 0 or 1 (clear or almost clear) or as a 75% reduction in Psoriasis Area and Severity Index (PASI).

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent.
* Subjects must be 18 years of age or older.
* Subject must be adult males or non-pregnant, non-lactating females.
* Female subjects of childbearing potential must state that they are using measures to avoid conception through active means including hormone replacement, intrauterine device, or abstinence.
* Subjects must be in general good health with no other skin disease, disease state or physical condition which would impair evaluation of psoriasis or which would increase their health risk by study participation.
* Subjects must be willing to receive an IM injection per protocol for 1 year.
* Must require systemic therapy or phototherapy for their psoriasis, as determined by the investigator prior to Visit 1. Objectively this equates to

Inclusion criteria of either:

* IGA≥3 on a 0-5 scale and BSA≥10%
* PASI ≥12

  * Subjects may not be taking any other systemic therapies or receiving phototherapy during the duration of the study. Subjects are required a 4 week washout period from any systemic medication or phototherapy prior to enrolling in the study and starting treatment with alefacept.
  * There is no washout for topical corticosteroid medications. Stable dosing of topical corticosteroids may be used up until the first dosing visit.

Exclusion Criteria:

* Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.
* Subjects have guttate, pustular, erythrodermic or rapidly flaring psoriasis.
* Current enrollment in any research study.
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within the 3 months prior to the first dose of investigational drug.
* Any subject who has a CD4<250 cells/µL at study entry.
* Treatment with another investigational drug or approved therapy within 28 days prior to study drug administration.
* Treatment with systemic retinoids, systemic steroids, methotrexate, cyclosporine, azathioprine, thioguanine, etanercept, efalizumab, infliximab, adalimumab or mofetil or other systemic immunosuppressant agents within the 28 days prior to investigational drug administration.
* Phototherapy, including Ultraviolet B (UVB) and Psoralen + Ultraviolet A (PUVA), within 28 days prior to investigational drug administration.
* Known HIV+, known viral Hepatitis infection, known tuberculosis infection.
* History of systemic malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feldman, MD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen subjects with moderate to severe chronic plaque type psoriasis were recruited from the Wake Forest University Health Sciences Dermatology Clinic
Groups:
- Alefacept: All subjects will receive 15 mg of alefacept IM per week (unless CD4<250 cells/µL, then dose will be withheld), for 16 weeks of treatment. After that they will be receive alefacept (15mg IM) once every 4 weeks for 8 months
Period: Overall Study
Arm/Group | Alefacept
Started | 15
Completed | 12
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Desired Alternate Therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alefacept
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Efficacy
Description: Efficacy of continuous use of alefacept as defined as the number of participants with a 75% reduction in Psoriasis Area and Severity Index (PASI) score from Baseline to week 52
Time Frame: 52 weeks
Measure: Number; unit: #Participants
Arm/Group | Alefacept
Number analyzed (Participants) | 15
#Participants | 1

2. Secondary Outcome: Safety of Alefacept Using CD4 Counts
Description: Number of participants experiencing CD4 cell counts below 250/uL
Time Frame: 52 weeks
Measure: Number; unit: Participants
Groups:
- Alefacept: All subjects received alefacept injections per FDA dosing guidelines for the duration of the 52 weeks study
Arm/Group | Alefacept
Number analyzed (Participants) | 15
Participants | 2

ADVERSE EVENTS:
Arm/Group | Alefacept
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alefacept (N=15)
Low CD4 cell count (Immune system disorders) | 1 (1) — CD4 cell count <250 cells/uL
Severe allergic contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alefacept (N=15)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Generalized itching (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No